CLINICAL TRIAL: NCT04714801
Title: A Danish, Single Centre, Double-blind, Randomized Study Evaluating Allogeneic Adipose Tissue Derived Mesenchymal Stromal Cell Therapy to Reduce Primary Graft Dysfunction After Lung Transplantation
Brief Title: Adipose Derived Mesenchymal Cell Treatment in Lungtransplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, JKastrup, MD professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC Lungtransplantation
Record Dates: First submitted 2020-05-29; First posted 2021-01-19 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Lung Transplant Rejection
Keywords: lung transplantation; Rejection; mesenchymal stromal cell; immune modulation; clinical trial; treatment
MeSH Terms: conditions — Rejection, Psychology | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled dose titrating study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infusion of 100 million ASC (Active Comparator): Infusion of 100 million adipose derived mesenchymal stromal cells from healthy donors
  Interventions: Drug: adipose derived mesenchymal stromal cells
- Infusion of 200 million ASC (Active Comparator): Infusion of 200 million adipose derived mesenchymal stromal cells from healthy donors
  Interventions: Drug: adipose derived mesenchymal stromal cells
- Infusion of placebo (Placebo Comparator): Infusion of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: adipose derived mesenchymal stromal cells — Intravenous infusion of cells
  Other Names: CSCC_ASC
  Arms: Infusion of 100 million ASC; Infusion of 200 million ASC
Drug: Saline — Intravenous infusion of saline
  Arms: Infusion of placebo

SUMMARY:
To investigate safety of treatment with allogeneic adipose tissue-derived mesenchymal stromal cells (ASCs) in patients undergoing lung transplantation, to evaluate whether the treatment can reduce host immunological reaction towards the graft, and to reduce the ischemic reperfusion-injury after transplantation.

DETAILED DESCRIPTION:
The emerging field of stem cell therapy holds promise of treating a variety of diseases. Especially the mesenchymal stromal cells from bone marrow (BMSCs) or adipose tissue (ASCs) have proven their potential for regenerative therapy in patients with ischemic heart disease. Both of these cell types have putative immunomodulatory properties, as they have demonstrated to actively suppress the immune system and hereby evade recognition.

This knowledge will be transferred into studies in the ischemic reperfusion-injury/primary lung graft dysfunction in lung transplantation, and in suppressing the initial host immunological response towards the transplanted lung where a high degree of immunological and inflammatory activity is involved.

We will conduct a clinical trial in which patients receiving lung transplantation will be randomized to either placebo or treatment with allogeneic MSCs from adipose tissue. The aim is to assess the impact of MSCs on primary graft dysfunction.

The perspective is that this new information can be of pivotal importance and potentially be a paradigm shift for the clinical problems seen in the first period after lung transplantation and reduce the long-term graft rejection and dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female lung recipients 18-70 years of age undergoing primary double (including size reduction) lung transplantation.
* Patient willing and capable of giving written informed consent for study participation and anticipated to be able to participate in the study for 3 months.

Exclusion Criteria:

* Recipients of multi-organ transplant, and or previously transplanted with any solid organ, including previous lung transplantation.
* Patients scheduled for single lung transplantation.
* Patients in need of acute transplantation e.g. patients on urgent call for transplantation and patients on respirator or on extra corporal membrane oxygenation (ECMO) treatment at time of transplantation.
* Patients that based on crossmatch prior to transplantation have need for additional immunosuppressive treatment
* Donor lung cold ischemic time > 12 hours.
* Patients with platelet count < 50,000/mm3 at the evaluation before transplantation.
* Patients who are unlikely to comply with the study requirements.
* Patient unable to participate in the study for the full study period
* Patients with any past (within the past 3-5 years) or present malignancy (other than excised basal cell carcinoma).
* Females capable of becoming pregnant must have a negative pregnancy test prior to transplantation. After inclusion, they must use contraceptives for 2 months following the given stem cell treatment. The pill, spiral, depot injection of progesterone, sub-dermal implantation, hormonal vaginal ring and transdermal patch regarded as safe contraceptives.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary graft dysfunction (PDG) | 3 days after treatment
  Difference in presence or not presence of Primary graft dysfunction (PGD) after transplantation in ASC treated patients compared to controls.
  Primary graft dysfunction is defined, according to the International Society for Heart and Lung Transplantation (ISHLT), as presence of both pulmonary infiltrates and hypoxemia occurring within the first 72 hours after transplantation

SECONDARY OUTCOMES:
Kidney glomerular Filtration Rate | 12 weeks after treatment
  Difference in estimated Glomerular Filtration Rate (eGFR)/1,73 m2. Normal > 60 ml/min
Inflammatory markers | through the 12 weeks
  Differences in C-reactive protein. Normal value < 10mg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, MD Professor, Study Director — Rigshospitalet, Denmark; Michael Perch, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- 2014 Department of Cardiology, The Heart Centre, University Hospital Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We are open for collaboration with external research groups, but have no presently plans
Supporting Information: Study Protocol, ICF
Time Frame: When the study is finalized and published
Access Criteria: Relevant documented use of data.

REFERENCES:
- [Derived] Qayyum AA, Lund TK, Jensen PB, Jensen K, Haack-Sorensen M, Ekblond A, Norgaard MJ, Moller-Sorensen H, Mathiasen AB, Moller CH, Rorvig SB, Kalhauge A, Bruunsgaard H, Litman T, Johansen EM, Hojgaard LD, Kastrup J, Perch M. Allogeneic mesenchymal stromal cell therapy on primary graft dysfunction after lung transplantation. JHLT Open. 2025 Mar 20;8:100254. doi: 10.1016/j.jhlto.2025.100254. eCollection 2025 May. PMID 40247997